CLINICAL TRIAL: NCT02394717
Title: Policy to Practice: Statewide Rollout of YMCA Childhood Obesity Standards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael Beets, Principal Investigator, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00031161; 1R01HD079422-01 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet, Healthy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Other): All YMCA programs will receive the Healthy Eating and Physical Activity Intervention throughout the study. All programs will receive the HEPA Strategies intervetion to assist them with achievement of the HEPA Standards.
  Interventions: Behavioral: Healthy Eating and Physical Activity

INTERVENTIONS:
Behavioral: Healthy Eating and Physical Activity — Create partnerships with ASPs to help facilitate changes in programming to meet the National Afterschool Alliance's HEPA Standards.
  Other Names: HEPA

SUMMARY:
The investigators long term-goal is to help YMCA programs across the nation successfully acheive the Y of USA "Healthy Eating and Physical Activity Standards". Our objective here is threefold. First, the investigators will work with South Carolina YMCA leadership to achieve the "Healthy Eating and Physical Activity Standards" and implement our HEPA Strategies in YMCA programs across the state, evaluate the uptake of and adherence to the standards and strategies, and identify factors that influence their implementation. Second, the investigators will evaluate the impact of acheiving the standards on children's MVPA and the serving and consumption of FV and water during the programs. Third, the investigators will evaluate the costs associated with and the cost-effectiveness of meeting the standards in terms of improvements in activity and healthy eating.

DETAILED DESCRIPTION:
The investigators research team developed a conceptual framework that identifies critical modifiable levers within Out of School Time programs that can be altered and/or strengthened to reach policy or standards goals. These include the policy environment at the national, state and local levels; characteristics of the individual site, program leadership, staff, and children; and existing outside organizational partnerships. This framework was informed by complex systems change, social ecology, systemic capacity building , and the literature on the impact of public health policy that identifies key elements of the system to be targeted as well as possible influences on those elements.

Viewing OST programs as complex systems, "Healthy Eating and Physical Activity Standards" represent one of many leverage points within a system. Existing efforts to implement standards rest solely upon the voluntary adoption of the standards, with little to no other changes to the OST program setting. It is clear from our preliminary work and comprehensive reviews that OST programs are falling short of meeting goals set forth in the standards.

ELIGIBILITY:
Inclusion Criteria:

* All children enrolled in participating afterschool programs will be eligible to take part in the study.

Exclusion Criteria:

* Any physical/orthopedic impairment that would limit a child's ability to participate in regular physical activity (e.g., wheelchair user).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2014-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in proportion of children meeting physical activity policy | Baseline, Fall of Year 2, and Fall of Year 3
  We will assess the number of children meeting the physical activity policy of 30 minutes or more of moderate-to-vigorous physical activity

SECONDARY OUTCOMES:
Changes in Nutritional Quality of Snacks | Baseline, Fall of Year 2 and Fall of Year 3
  We will assess quality of snacks served at the ASPs in terms of number of fruits and vegetables served per week.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Beets, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Beets MW, Glenn Weaver R, Brazendale K, Turner-McGrievy G, Saunders RP, Moore JB, Webster C, Khan M, Beighle A. Statewide dissemination and implementation of physical activity standards in afterschool programs: two-year results. BMC Public Health. 2018 Jul 3;18(1):819. doi: 10.1186/s12889-018-5737-6. PMID 29970046